CLINICAL TRIAL: NCT06172816
Title: The Second Affiliated Hospital of Chongqing Medical University
Brief Title: A Cohort Study on the Clinical Characteristics and Prognosis of HIV/AIDS Patients Infected With SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023IITxG12
Record Dates: First submitted 2023-12-10; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-01

CONDITIONS: PLWH; Covid-19; Clinical Features; Prognosis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLWH: the people living with HIV
  Interventions: Other: SARS-CoV-2
- HC: the people without disease
  Interventions: Other: SARS-CoV-2

INTERVENTIONS:
Other: SARS-CoV-2 — a virus infection

SUMMARY:
On February 11th, 2020, the International Classification of Viruses named the disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) as novel coronavirus (COVID-19, Covid-19 for short). At present, COVID-19 has become a global pandemic. However, the persistent replication of HIV in PLWH and the cellular immunodeficiency and persistent inflammation caused by it may have different effects on the susceptibility, severity and course of Covid-19. Several large cohort studies have found evidence of increased risk of hospitalization and death in patients with HIV and Covid-19 co-infection. Meanwhile, a meta-analysis of 22 studies shows that HIV infection is still an important risk factor for acquiring Covid-19 infection, and it is associated with a higher risk of death in COVID-19. In order to further clarify the clinical features and prognosis of HIV co-infection with Covid-19 and explore its immune mechanism, so we will carry out the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old; Patients diagnosed with HIV in accordance with the Chinese AIDS Diagnosis and Treatment Guidelines.

Exclusion Criteria:

* Hypertension, diabetes and other metabolic related diseases; Severe circulatory and respiratory diseases; Patients with immune-related diseases and immunosuppressants; Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people and people living with HIV which is immunodeficient.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical features and prognosis | 2022.11-2023.1
  the clinical features and prognosis between healthy people and PLWH infected with Omicron
antibody titer | 2022.11-2023.1
  the SARS-CoV-2 specific antibody titers between healthy people and PLWH infected with Omicron

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality, China